CLINICAL TRIAL: NCT03008824
Title: Micronutrients in Pregnancy as a Risk Factor for Diabetes and Effects on Mother and Baby: PRiDE Study
Brief Title: Micronutrients in Pregnancy as a Risk Factor for Diabetes and Effects on Mother and Baby
Acronym: PRiDE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Warwick (Other)
Collaborators: George Eliot Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Dr P Saravanan, Associate Clinical Professor, University of Warwick
Other Study IDs: MR/J000094/1
Record Dates: First submitted 2016-12-22; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum and whole blood for isolating DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
There is a rapidly escalating epidemic of obesity and type 2 diabetes across the world, with the fastest rise occurring in low- and middle-income countries. India not only has one of the highest rates in the world, but the disease starts at a younger age and lower levels of body weight than in UK white caucasians. Among city-dwelling Indians, approximately 8% of people aged 30-40 years already have diabetes. This is creating a heavy burden of disease and disability, and an intolerable economic burden through medical costs and lost earnings. Until now, efforts to prevent diabetes have mainly focussed on modifying the diet, lifestyle and activity of at-risk adults (for example those who are overweight, have a family history of diabetes or already have high blood sugar). However, recent research has indicated that factors acting in early life (during development in the womb) place an individual at risk of later diabetes. These include maternal malnutrition and low birthweight, and diabetes in the mother during pregnancy. Our research has shown that Indian mothers often have low vitamin B12 levels, which in turn causes high blood levels of a harmful metabolite (homocysteine). We have shown that these mothers get more diabetes in pregnancy. Their children are more likely to born with a low birth weight, and develop more body fat and higher plasma insulin levels during childhood, which are signs of higher diabetes risk in later life. The risk is increased further if the mother has normal or high status for another B vitamin, folate. Thus, we have shown, for the first time a link between a specific nutritional deficiency in the mother and diabetes risk in the next generation. One possible mechanism for the effect of maternal nutrition on risk of diabetes in her children is through epigenetic effects, whereby the nutritional environment during early development affects the switches that control gene expression. Since these switches are passed on via either parent, we think it is possible that paternal vitamin B12 status could also be important.

DETAILED DESCRIPTION:
Background:

Risk of GDM and offspring's metabolic risk:

There is an escalating epidemic of type 2 diabetes (T2D) across the world in all ethnic groups, in particular, people of South Asian origin. Current strategies for preventing T2D rely mainly on altering risk factors such as obesity, sedentary lifestyle and healthy eating. Though this is important, it is unlikely to make a big impact on this escalating epidemic, which consumes significant proportion of health care budgets, world-wide. Some of the risk of developing metabolic diseases such as T2D and cardiovascular disorders (CVD) are evident even at birth. Indeed, recent research suggests that factors acting during early development, including foetal growth restriction and exposure to gestational diabetes (GDM) in the mother increases diabetes and obesity risk in later life. The investigators recent work has shown that maternal vitamin B12 insufficiency and hyper-homocysteinaemia, in combination with normal/high maternal folate status, is associated with an increased risk of GDM in the mothers, growth restriction in the foetus, and adiposity and insulin resistance in the children.

GDM is described as glucose intolerance first recognised in pregnancy. Similar to T2D, GDM is also increasing at an alarming rate, attributed partly to increasing maternal age and body weight. The current estimate is around 4% of all pregnancy though this could increase to as much as 17% if the new IADPSG guidelines are implemented. Women who develop GDM are at 7-8 times higher risk of T2D13 and the children born to them are at higher risk of developing T2D, abdominal obesity and metabolic syndrome later in life thus increasing their risk of CVD in adulthood. Though the exact etiological processes of such increased risk not clear, some of these effects could act through epigenetic mechanisms (intra-uterine programming).

The study by Krishnaveni et al raises an intriguing possibility for a simple measure for preventing GDM and future T2D. It is believed that the high prevalence of B12 insufficiency in India was attributed to vegetarianism. As the majority of the UK population is non-vegetarian, it is conceivable that B12 deficiency is unlikely during pregnancy. However, the investigators have recently shown: a) B12 deficiency is not uncommon in women of childbearing age (14%) and pregnant women (20% at 16-18 weeks of pregnancy) and b) B12 deficiency in GDM is associated with higher BMI and higher birth weight in a clinic population.

Psychological impact of GDM:

Mothers who are screened for GDM have lower perceived well-being. Diagnosis of GDM during pregnancy often comes as a shock and causes significant distress to expectant mothers. There is some evidence that such distress improves after treatment, presumably due to education and support. These limited data come from women of Caucasian origin and no such data exists in women of South Asian origin.

To confirm these observations in the UK multi-ethnic population, the investigators plan to carry out an adequately powered case-control study to examine: a) the influence of early pregnancy B12, folate and homocysteine levels (as well as other clinical, biochemical and genetic markers) on the risk of GDM and offspring's risk of future metabolic disorders by measuring detailed anthropometry of the babies along with their biochemical and genetic markers from the cord blood; and b) the psychological impact of diagnosis of GDM by measuring the anxiety and distress by questionnaires.

Hypothesis:

Imbalance of B12, folate and homocysteine in early pregnancy predicts the risk of GDM in mothers and metabolic risk of offspring

Research plan and methodology:

Population: Pregnant women attending antenatal care in the UK; Cases will be pregnant women carrying singleton foetuses, without pre-gestational diabetes, who are diagnosed with GDM during the pregnancy. Equal number of South Asian and Caucasian mothers with GDM will be recruited.

Intervention / Exposure: Maternal vitamin B12, folate and homocysteine levels in early pregnancy (<16 weeks of gestation) Comparison Group: Mothers from the cohort who do not develop GDM and are matched in age, parity and BMI to the cases

Study Design:

A prospective observational case-control study designed to compare early pregnancy B12, folate and homocysteine levels in pregnant women who develop GDM (cases) and those who do not (controls).

Sample size:

There is no published data on the rate of B12 deficiency in GDM women in the UK and limited data exists in non-GDM women in Caucasians. Preliminary results from the investigators' group have shown that approximately 15% insufficiency in non-GDM and around 20%-25% in GDM women of Caucasian origin. To detect a 5% difference in the prevalence of B12 insufficiency with 90% power at the 5% significance level, 700 GDMs will be required. We plan to identify 1400 controls matched for age, BMI and parity. To achieve this,4080 pregnant women will be required in their first trimester over the 2.5 years (if 20% develop GDM). Allowing for a 10% drop-out rate and for age, parity & BMI matching 4500 pregnant mothers will be recruited.

Implementation plan:

Several study launches are planned to raise the awareness among the public, midwifes and general practitioners in the region. The relevant clinical research networks (CRNs) will be involved from the beginning both to raise the awareness and for direct involvement in the study.

Most potential participants will be given the participant information sheet (PIS) when they are seen for their booking visit by the community midwife. The midwife will assess their eligibility for the study and hand out the PIS if they fit the inclusion criteria. The midwife will inform the research team of the mothers' details via a Reply Slip if she has no objection to be contacted. The research team will then contact the mother and if possible, the recruitment visit will be planned to coincide with her booking bloods or dating scan appointment (usually around 12 weeks of gestation) to minimise the study visits ('Research Team Recruitment', see right-hand side of Recruitment Flow chart).

In the situation where a mother has been identified by her midwife as fitting the inclusion criteria for the study (i.e. she has high-risk factors for GDM and is therefore referred for a GTT), but is not given a PIS at the booking visit, the research team will send this out by post to the mother with an invitation letter.

Feedback from the mothers at the recruitment visit (i.e. dating scan) suggests that the mothers would have been happy to partake in the study at the same visit as receiving the PIS for 4 main reasons: 1) the study (and the PIS) is simple to understand; 2) they spend a significant amount of time awaiting scan and midwife appointment during this visit; 3) they want to have their blood sample taken at the same visit (mothers have a blood test routinely as a standard care); and 4) they prefer not to come back for a separate visit. The investigators also believe this is reasonable as this is a non-interventional study and provides opportunity for more mothers to participate in the study. Therefore if the mother has had enough time to read and understand the PIS and provides consent, she could be recruited straightaway and blood tests done together with her routine bloods on the same day. However, if she prefers to take the PIS away and have more time to decide, the research team will see her at a future date. Such a strategy can also be replicated in the community booking visit to facilitate participation in the study.

The participants will have basic demographic information collected and anthropometric measurements done during the recruitment visit and be asked to fill out physical activity and psychological well-being questionnaires. To facilitate the ease of filling the questionnaire, where ever possible patients will be given iPads to complete them. We will then collect blood samples (approximately 15-20ml in addition to their routine booking bloods), a urine and stool sample (optional) from them.

Mothers will have their OGTT at 24-28 weeks gestation and further blood, urine and stool (optional) samples will be taken at this time for study purposes. Modified WHO (1998) and NICE criteria will be used to diagnose gestational diabetes or not(i.e. fasting plasma glucose ≥ 6.1 mmol/l OR fasting plasma glucose < 6.1 mmol/l and 2 hour plasma glucose > 7.8mmol/l but < 11.1 mmol/l on 75g glucose tolerance test). The criteria will be changed if the new IADPSG criteria is adopted during the course of the study (or NICE updates its criteria). The mothers will be asked to fill out further psychological well-being questionnaires during the waiting time during the OGTT and for mothers subsequently diagnosed with GDM, when they attend the antenatal-diabetes clinic.

The remainder of a participant's antenatal care will then carry on in the joint antenatal-diabetes clinic (if she has been diagnosed with GDM) or in the community (for non-GDM mothers, unless she has any other indication to be referred to the obstetric clinic).

All the participants will have their deliveries in one of the NHS Hospitals involved in the study. Cord blood, a piece of cord and placental biopsies (around 2cm each) will be taken at the time of birth as well as detailed birth and neonatal outcome data and a stool sample from the baby shortly afterwards. Baby's body fat content and distribution will be measured by the 'PEAPOD' machine. This is a non invasive, baby friendly way of accurately measuring the fat distribution in the baby. This is optional. For mothers who have Caesarean sections (for medical/obstetric reasons), we will ask for separate consent to take a sample of abdominal fat and subcutaneous as well as myometrial smooth muscle tissues. All the samples obtained will stored for future DNA isolation.

During the post-natal OGTT for GDM mothers (6 weeks post-partum) additional blood samples will be collected and stored. Also, well-being questionnaires will be given out to all participants post-natally. From 3 to 12 months, breast feeding mothers will be contacted either through postal questionnaire or over the telephone.

Appendices and summary of additional data collection:

1. IPAQ (Physical activity) questionnaire - baseline
2. PhQ9 questionnaire - at baseline
3. GAD7 questionnaire - at baseline
4. Warwick - Edinburgh well being questionnaire (WEMWBS) - baseline, 24-28 weeks and 6 weeks postpartum during OGTT
5. Euro-QoL - Quality of Life measure at baseline, 24-28 weeks and 6 weeks postpartum GTT
6. Socio-economic measure - baseline, 24-28 weeks and 6 weeks postpartum GTT
7. PSQI (Pittsburgh Sleep Quality Index questionnaire)
8. Breast feeding questionnaire (post natal)

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women <16 years of age
* High risk for GDM (at least 1 of the risk factors) - BMI >30
* Previous GDM
* First degree relatives with GDM
* Previous unexplained still birth
* Previous baby >4.5kg
* PCOS
* Ethnic minority groups
* Age >35years

Exclusion Criteria:

* Pregestational Type 1 or Type 2 Diabetes
* Diagnosis of B12 or folate deficiency in the current pregnancy
* Previous pregnancies with NTDs
* Diagnosis of severe aneamia (<10g/dL)
* Vitamin B12 injections in the previous 6 months

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All pregnant women between 18-75 years of age who satisfy NICE criteria for GDM screening
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2012-09; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Differences in B12 levels between GDM and Controls | 5 Years

SECONDARY OUTCOMES:
Differences in B12 levels in South Asians and White Caucasians | 5 years
Differences between offspring birth weight between GDM and controls | 5 years
Differences between offspring adiposity between GDM and controls | 5 years
Differences between offspring birth weight between South Asians and White Caucasians | 5 years
Differences between offspring adiposity between South Asians and White Caucasians | 5 years
Clinical and Biochemical predictors of GDM in the first trimester | 5 years
Predictors of abnormal post-natal OGTT in the first trimester | 5.5 years

OTHER OUTCOMES:
Psychological impact of the diagnosis of GDM in each ethnicity | 5 years
Role of sedentary behavior on incident GDM | 5 years
Role of physical activity on incident GDM | 5 years
Role of maternal 1-C metabolites on incident GDM | 5 years
Role of maternal 1-C metabolites on metabolic risk in the offspring at birth | 5 years
Role of maternal metabolic risk factors on offspring adiposity measured by PEAPOD | 8 years
Validation of newborn adiposity measured by skin-fold thickness and objective measurement by PEAPOD | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Ponnusamy Saravanan, FRCP PhD, Principal Investigator — University of Warwick
Locations (1):
- University of Warwick, Coventry, Coventry, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
A core dataset and the metatdata that is funded by MRC will be archived

REFERENCES:
- [Derived] Saravanan P, Sukumar N, Adaikalakoteswari A, Goljan I, Venkataraman H, Gopinath A, Bagias C, Yajnik CS, Stallard N, Ghebremichael-Weldeselassie Y, Fall CHD. Association of maternal vitamin B12 and folate levels in early pregnancy with gestational diabetes: a prospective UK cohort study (PRiDE study). Diabetologia. 2021 Oct;64(10):2170-2182. doi: 10.1007/s00125-021-05510-7. Epub 2021 Jul 22. PMID 34296321